CLINICAL TRIAL: NCT02083588
Title: A Prospective Trial to Explore the Efficacy of the H1-Coil Deep Transcranial Magnetic Stimulation (TMS) in Subjects With Fibromyalgia
Brief Title: A Prospective Trial to Explore the Efficacy of dTMS in Subjects With Fibromyalgia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shalvata Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FMS_01
Record Dates: First submitted 2014-02-26; First posted 2014-03-11 (Estimated); Last update posted 2014-03-11 (Estimated); Status verified 2014-03

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; dTMS; pain; PFC; Subjects with Fibromyalgia
MeSH Terms: conditions — Fibromyalgia; Pain

ARMS (1):
- open - single arm (Experimental): All subjects will receive prefrontal deep rTMS of H1 Coil (75 trains of 2 seconds, 20 Hz, with 20 seconds inter-train intervals, up to 120% of motor threshold, a total of 3000 pulses per session), for 4 weeks, 5 days a week, overall 20 sessions.
  Interventions: Device: dTMS

INTERVENTIONS:
Device: dTMS — All subjects will receive prefrontal deep rTMS of H1 Coil (75 trains of 2 seconds, 20 Hz, with 20 seconds inter-train intervals, up to 120% of motor threshold, a total of 3000 pulses per session), for 4 weeks, 5 days a week, overall 20 sessions.
  Other Names: The Brainsway Ltd. H1-Coil

SUMMARY:
Fibromyalgia Syndrome (FMS) is a highly prevalent condition often affecting individuals in the prime of life, causing severe reduction in quality of life and productivity, as well as social isolation, anxiety, and depression. The purpose of this study is to explore the efficacy of H1 deep TMS for the treatment of FMS patients. In addition, the investigators attempt to assess the effect of dTMS on the perception and modulation of pain in patients suffering from FMS.

DETAILED DESCRIPTION:
Fibromyalgia Syndrome (FMS) is a highly prevalent condition often affecting individuals in the prime of life, causing severe reduction in quality of life and productivity, as well as social isolation, anxiety, and depression. FMS has recently been estimated to affect approximately 2.6% of the Israeli population. Over the last decade, it has repeatedly been shown that Transcranial Magnetic Stimulation (TMS) of the primary motor cortex (M1) induces an analgesic effect both in experimental pain, as well as in various chronic pain conditions, possibly by activating intrinsic pain-modulation systems.

Thus, the purpose of this study is to explore the efficacy of H1 deep TMS for the treatment of FMS patients. In addition, the investigators attempt to assess the effect of dTMS on the perception and modulation of pain in patients suffering from FMS.

The study will take place in Shalvata Mental Health Center, After receiving the hospital's BRI approval. Forty FMS patients between 18-65 years of age will sign an informed consent form, and be randomized to an active arm (dTMS) and a placebo arm (sham-dTMS). Twenty treatments will be delivered to each subject over a period of 4 weeks. At base-line subjects will complete a series of epidemiological and clinical questionnaires (assessing symptoms of FMS, depression, pain, anxiety), as well as pain sensation and modulation tests. At the termination of the study and two weeks after the final treatment all questionnaires and physical measurements will be re-administered for a final assessment of post-treatment status comparison with initial status The importance of the study lies in its potential to: 1) provide evidence for the efficacy of dTMS in treating patients suffering from FMS 2)enhance the investigators understanding of the pathophysiology of FMS and its underlying pain perception and modulation mechanisms 3) explore the role of the Dorso-Lateral-Prefrontal-Cortex (DLPC) in modulating pain and as a possible target to further therapeutic interventions in FMS.

ELIGIBILITY:
Inclusion Criteria:

* Concomitant medication for pain and sleep disorders will be allowed provided the dose administered had been stable for at least 2 months before enrollment and remains stable throughout the study.
* Gave informed consent for participation in the study.

Exclusion Criteria:

* Subjects will be excluded if evidence is found of inflammatory rheumatic disease, autoimmune disease, or other painful disorders that might confound assessment of FMS pain.
* Subjects diagnosed with a current primary psychiatric condition - including major depression or major personality disorders according to Diagnostic and Statistical Manual of Mental Disorders-IV criteria - or a history of substance abuse will be excluded, as well as pregnant subjects.
* History of any metal in the head (outside the mouth).
* Known history of any metallic particles in the eye, implanted cardiac pacemaker or any intracardiac lines, implanted neurostimulators, surgical clips or any medical pumps.
* History of head injury.
* History of seizure or heat convulsion.
* History of epilepsy or seizure in first degree relatives.
* History of frequent or severe headaches.
* Use of hearing aids for hearing loss.
* Known history of cochlear implants.
* History of drug abuse or alcoholism during the last year.
* Serious and unstable medical condition, which is likely to exacerbate or endanger the patient during the treatment period.
* Inadequate communication with the patient.
* Subjects declared as legally incompetent, with an appointed physical guardian and/or cannot sign informed consent due to cognitive incompetence.
* Participation in current clinical study or clinical study within 30 days prior to this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-03; Primary Completion 2015-03 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
pain intensity - past 24h | at baseline, and after treatment number 5, 10, 15 and 20, in addition to a final examination on follow up (two weeks after determination).
  Change in self-reported average pain intensity over the last 24 hours will be measured at the end point with the numerical scale (0 = no pain, 10 = maximal pain imaginable) of the VAS-FIQ.

SECONDARY OUTCOMES:
pain dimensions | baseline and follow up (two weeks after determination of treatment).
  1. Change of sensory and affective pain dimensions will be measured at the end point using the McGill Pain Questionnaire.
  2. Change of the impact of pain and FMS on quality of life, will be measured at the end point using the BPI items for pain interference.
  3. change of sensitivity to painful stimuli will be evaluated by physical measurements:
     * mechanical Temporal Summation - mTS
     * Sensory threshold
     * Thermal Pain Threshold
     * CPM
     * WPI
     * SSS

CONTACTS AND LOCATIONS:
Locations (1):
- Shalvata MHC, Hod Ha-sharon, Israel